CLINICAL TRIAL: NCT00939380
Title: Facilitating Parent Adaptation to Pediatric Transplant: The P-SCIP Trial
Acronym: P-SCIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Hospital Los Angeles (Other); Columbia University (Other); Emory University (Other); Memorial Sloan Kettering Cancer Center (Other); University of Medicine and Dentistry of New Jersey (Other); Icahn School of Medicine at Mount Sinai (Other); Weill Medical College of Cornell University (Other); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 130906; 1R01CA127488-01A1 (NIH); CDR0000632012 (Registry Identifier: PDQ (Physician Data Query)); FCCC-07848; 0220090280 (Other: IRB Number); P30CA072720 (NIH); IRB#07-848; 15032-01 (Other: Fox Chase number); NCT00953082 (obsolete NCT alias)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Childhood Cancers
Keywords: hematopoietic stem cell transplant; bone marrow transplant; children; parents; counseling; depression
MeSH Terms: conditions — Depression | interventions — CD-ROM; Respite Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- P-SCIP (Experimental): Arm I (Parent Social-Cognitive Intervention Program [P-SCIP]): Participants undergo five 60-minute behavioral intervention sessions once or twice weekly for 3 weeks to learn how to engage in effective social and cognitive processing to deal with fears and worries about the transplant and transplant-related concerns. Participants receive a laptop computer and a CD-ROM after the first session.
  Interventions: Behavioral: Behavioral intervention sessions; Other: CD-ROM
- BPC (Experimental): Arm II (Best-recommended Psychosocial Care [BPC]): Participants undergo usual care and receive a "Discovery to Recovery" DVD and pamphlet developed by the National Marrow Donor Program (NMDP) describing psychological issues associated with hematopoietic stem cell transplantation (HSCT), the booklet "Top Tips for Parent Caregivers During the BMT Process" published by National Marrow Donor Program-Link describing caregiver issues during HSCT and advice on how to handle them, 2 walkie-talkies, a laptop to view the DVD, and 5 hours of respite care from a child-life specialist once or twice weekly for 3 weeks.
  Interventions: Other: DVD and pamphlet; Other: Respite care

INTERVENTIONS:
Behavioral: Behavioral intervention sessions — Participants undergo five 60-minute behavioral intervention sessions once or twice weekly for 3 weeks to learn how to engage in effective social and cognitive processing to deal with fears and worries about the transplant and transplant-related concerns.
  Arms: P-SCIP
Other: CD-ROM — Participants receive a laptop computer and a CD-ROM after the first session of behavioral intervention.
  Arms: P-SCIP
Other: DVD and pamphlet — Participants receive a "Discovery to Recovery" DVD and pamphlet developed by the National Marrow Donor Program (NMDP) describing psychological issues associated with hematopoietic stem cell transplantation (HSCT), the booklet "Top Tips for Parent Caregivers During the BMT Process" published by National Marrow Donor Program-Link describing caregiver issues during HSCT and advice on how to handle them, 2 walkie-talkies, a laptop to view the DVD.
  Arms: BPC
Other: Respite care — Participants receive 5 hours of respite care from a child-life specialist once or twice weekly for 3 weeks.
  Arms: BPC

SUMMARY:
The investigators have developed a parent social-cognitive processing intervention (P-SCIP) to help decrease distress among parent caregivers of children undergoing hematopoietic stem cell transplant (HSCT). The investigators will evaluate the efficacy of P-SCIP in reducing short- and long-term distress and parenting stress among 300 parents of children undergoing HSCT. P-SCIP will be delivered during the child's inpatient HSCT hospitalization and is specifically designed to improve parent social (e.g., sharing concerns) and cognitive (e.g., acceptance) processing of the transplant experience. The intervention includes five in-person sessions that are accompanied by an interactive CD-ROM. The CD-ROM complements the materials in the in-person sessions and provides parents with the opportunity to enhance and deepen their cognitive and social processing of the HSCT experience. The intervention will be tested against best-practices psychosocial care (BPC) available in four enriched pediatric HSCT settings across the United States. P-SCIP will be provided to both Spanish- and English-speaking parents. Participants will complete measures of psychological distress, well-being, and social and cognitive processing at the time of HSCT, two, six and twelve months after HSCT. Research questions will address the effects of P-SCIP versus BPC on parent psychological adaptation and social and cognitive processing, as well as evaluate parent personal resources as well as child medical course variables that contribute to intervention response. The investigators will also examine barriers to participation in the intervention by comparing barriers to participation among parents who refuse participation in the trial and parents who accept.

ELIGIBILITY:
Inclusion Criteria:

* biological or foster parent of children under 19 years of age who are scheduled for HSCT within the next month
* participant is the primary caregiver
* participant must have phone service
* caregiver speaks, reads, and writes English or Spanish (Spanish is for Childrens Hospital Los Angeles and Columbia University only)

Exclusion Criteria:

* pediatric patient has a diagnosis of medulloblastoma or other cancer of the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2010-05; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 7 years
Beck Anxiety Inventory | 7 years
Mental Health Inventory | 7 years
Impact of Events Scale-Revised | 7 years
Axis I Structured Clinical Interview for DSM-IV (SCID) | 7 years

SECONDARY OUTCOMES:
Fear Structure | 7 years
Brief COPE | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Manne, Ph.D., Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (5):
- United States (5):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Emory University/Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York